CLINICAL TRIAL: NCT02299063
Title: The Protective Effect of the α2-agonist Dexmedetomidine on Mitochondrial Structure and Function for Children With Non-cyanotic Congenital Heart Defects Having Cardiac Surgery: A Randomized Controlled Trial.
Brief Title: Dexmedetomidine Effect on Mitochondrial Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, James O'Leary, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000044746
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Complication of Anesthesia; Ischaemia-reperfusion Injury
Keywords: Mitochondria; Dexmedetomidine; Heart Defects, Congenital
MeSH Terms: conditions — Reperfusion Injury; Heart Defects, Congenital | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (0.9% Saline) (Placebo Comparator): 0.9% Saline: bolus dose of 0.125mL/kg infused over 10 minutes, followed by a continuous infusion (CI) dose at 0.15mL/kg/hr for the duration of surgery.
  Interventions: Drug: 0.9% NaCl
- Dexmedetomidine (Experimental): Dexmedetomidine: bolus dose of 0.5 mcg/kg infused over 10 minutes, followed by a continuous infusion (CI) dose at 0.6 mcg/kg/hr for the duration of surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — A bolus dose of 0.5 mcg/kg infused over 10 minutes will be administered, followed by a continuous infusion for the duration of the surgery at 0.6 mcg/kg/hr.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: 0.9% NaCl
  Other Names: Normal Saline
  Arms: Placebo (0.9% Saline)

SUMMARY:
The investigators hypothesize that in addition to a known sympatholytic effect, intraoperative dexmedetomidine reduces adverse changes in mitochondrial function and structure attenuating ischaemia-reperfusion and end-organ injury for children with non cyanotic congenital heart defects having corrective heart surgery.

DETAILED DESCRIPTION:
PICO: For children with non cyanotic congenital heart defects having corrective heart surgery (P) does intraoperative dexmedetomidine (I) reduce real-time changes in mitochondrial function and content (O) compared with children not receiving dexmedetomidine (C).

The study drug (dexmedetomidine or placebo) will be mixed in a standardized syringe of 4mcg/mL for active syringes or 50mL 0.9% sodium chloride for placebo. Blinded syringes will be prepared by the Research Support Pharmacy.

Administration is via the existing central venous line. A bolus dose of 0.125mL/kg (0.5 mcg/kg dexmedetomidine) infused over 10 minutes will be administered, followed by a continuous infusion for the duration of the surgery. The dexmedetomidine/placebo continuous infusion (CI) dose will run at 0.15mL/kg/hr (0.6 mcg/kg/hr dexmedetomidine).

Blood samples will be obtained from each child at three points in the operating room: 1) after the induction of anesthesia, 2) at the first separation from CPB (prior to administration of blood products), and 3) at the end of the surgery.

Samples obtained will be analyzed for mitochondrial function and morphology, total cellular mitochondrial biomass, and mitochondrial deoxyribonucleic acid (mtDNA) damage:

1. After isolating lymphocytes, we will use high content imaging (HCI) to assess mitochondrial function and morphology. The lymphocytes will be stained with tetramethylrhodamine methyl ester (TMRM), which stains mitochondria in proportion to mitochondrial membrane potential, giving a metric for mitochondrial function. In addition, the cells will be stained with MitoTracker Green®, which can be used to assess mitochondrial morphology. Mitochondrial morphology will be quantified in a non-biased fashion using a mathematical image analysis algorithm.
2. After extraction of genomic DNA, total cellular mitochondrial biomass and mitochondrial DNA damage will be measured using traditional and long-patch quantitative polymerase chain reaction (PCR).

Myocardial tissue will be also collected prior to closure of the atriotomy. Samples will be placed into 3% buffered glutaraldehyde at the time of biopsy, and imaging of mitochondrial structure using electron microscopy will be performed.

ELIGIBILITY:
Inclusion Criteria:

* aged between 3 - 36 months
* having primary corrective heart surgery

Exclusion Criteria:

* recent surgery (< 3 months)
* previous chemotherapy
* previous transfusion of blood products
* neurodevelopmental disorders (including Trisomy 21)
* supplemental oxygen requirement (< 3 months)
* asthma requiring regular therapy
* obstructive sleep apnea
* the presence of concurrent infection or inflammation
* a known allergy to dexmedetomidine hydrochloride

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function (use high content imaging (HCI) | Intraoperative
  The primary outcomes for mitochondria will be grouped into mitochondrial function, morphology, content and mtDNA damage.

SECONDARY OUTCOMES:
Creatinine level (Marker of acute renal injury) | Postoperative day 1
  Marker of acute renal injury
Cardiac function (Left ventricular ejection fraction measured by trans-thoracic echocardiography) | Postoperative day 1
  Left ventricular ejection fraction measured by trans-thoracic echocardiography
Inotropes and vasopressors (Duration and dose of inotropes and vasopressors after surgery) | Postoperative day 1
  Duration and dose of inotropes and vasopressors after surgery

OTHER OUTCOMES:
Analgesic effects (Morphine equivalent dose of narcotics consumed) | Perioperative (from induction of anesthesia for 24 hours)
  Morphine equivalent dose of narcotics consumed
Sedative effects (Duration of intubation) | Perioperative (from induction of anesthesia for 24 hours)
  Duration of intubation.

CONTACTS AND LOCATIONS:
Overall Officials: James D O'Leary, MBBCh, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No